CLINICAL TRIAL: NCT00442312
Title: An Open Label,Switch Study of the Safety and Efficacy of Combigan Ophthalmic Solution(Brimonidine 0.2% and Timolol 0.5%)With Latanoprost Compared With Latanoprost Monotherapy in Patient With Glaucoma or Ocular Hypertension.
Brief Title: Combigan Ophthalmic Solution(Brimonidine 0.2% and Timolol 0.5%)With Latanoprost Compared With Latanoprost Monotherapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Genovate Biotechnology Co., Ltd., (Industry)
Collaborators: Allergan Medical (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: COM 003
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Glaucoma
Keywords: Combigan
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Combigan Ophthalmic Solutiom

SUMMARY:
This study is to evaluate the efficacy and safety of Combigan ophthalmic solution in combination with Latanoprost when the therapy is swiched from Latanoprost monotherapy in patient with Glaucoma or ocular hypertension.

Hypothesis:

1. Combigan Ophthalmic Solution provides addition IOP loweringwhen combined with Latanoprost.
2. The treatment with Combigan Ophthalmic Solution has an acceptable safety profile, as measured by ocular and systemic safety parameters.

DETAILED DESCRIPTION:
The purpose of this study is to comparethe efficacy and safety Ophthalmic Solution in combination with Latanoprost when the therapy is swiched from Latanoprost monotherapy in patient with Glaucoma or ocular hypertension.

The study will be open label, prospective, multi-centered where patients will be swiched from Latanoprostmonotherapy to a combination therapy of Latanoprost with Combigan Ophthalmic Solution.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, of legal age of consent.
2. Diagnosis of ocular hypertension (OHT) or glaucoma (incl. open angle glaucoma, chronic angle closure glaucoma, exfoliative glaucoma, pigmentary glaucoma or pseudophakic glaucoma) and requiring administration of IOP lowering eye drops.
3. Written informed consent has been obtained.
4. The patient can understand all study instructions, and is willing and able to comply with the schedule of visits and treatment.
5. Patient has been administering latanoprost eye drops as monotherapy in affected eye(s) for at least 12 weeks according to the approved product labeling.
6. Patient's Day 0 IOP > 18 mm Hg in the proposed study eye/s on established latanoprost therapy.
7. Patients who have used COMBIGAN® Ophthalmic Solution in the past must not have been discontinued from using this medication due to adverse events or due to lack of efficacy.
8. Day 0: negative urine pregnancy test for females of childbearing potential.

Exclusion Criteria:

1. .Uncontrolled systemic disease (e.g., hypertension, diabetes).
2. .Females who are pregnant, nursing, or planning a pregnancy, or females of childbearing potential who are not using a reliable means of contraception. A female is considered of child-bearing potential unless she is post-menopausal, without a uterus and/or both ovaries, or has a tubal-ligation.
3. .Known allergy or hypersensitivity to the study medication or components.
4. .Anticipated alteration of existing chronic therapy with agents which could have a substantial effect on IOP (including, but not necessarily limited to systemic adrenergic agents including beta-adrenergic blocking agents [e.g., propanolol, metoprolol, nadolol, timolol and atenolol]), substantial interaction with study medications, or interaction with study outcomes.
5. .Corneal abnormalities that would preclude accurate IOP readings with an applanation tonometer.
6. .Any other active ocular disease other than glaucoma or ocular hypertension (e.g., uveitis, ocular infections, or severe dry eye). However, patients with chronic mild blepharitis, cataract, age-related macular degeneration, or a background diabetic retinopathy can be enrolled at the discretion of the investigator.
7. .Required chronic use of other ocular medications during the study other than the study medications. Occasional use of artificial tears or topical decongestants and/or antihistamine is acceptable. Use of these within 24 hours of a scheduled study visit is prohibited.
8. .Ocular surgery within the past 3 months.
9. .Current enrolment in an investigational drug or device study or participation in such a study within 30 days of entry into this study.
10. .Patient has a condition or is in a situation which in the investigator's opinion may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study,
11. .Day 0 - Significant ocular irritation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43
Dates: Start 2006-05; Study Completion 2006-11

PRIMARY OUTCOMES:
The change of IntraOcular Pressure From baseline to week 12

SECONDARY OUTCOMES:
The change of IntraOcular Pressure on week 8.
The change of IntraOcular Pressure on week 12

CONTACTS AND LOCATIONS:
Overall Officials: Da-Wen Lu, Principal Investigator — Tri-Service General Hospital, Taiwan ROC
Locations (1):
- Allergan, Taipei, Taipei, Taiwan